CLINICAL TRIAL: NCT01893606
Title: Multicenter Randomized Withdrawal Clinical Trials of N-acetyl Glucosamine Capsule for Irritable Bowel Syndrome With Diarrhea (IBS-D) Treatment
Brief Title: Multicenter Withdrawal Clinical Trials of N-acetyl Glucosamine Capsule for IBS-D Treatment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Liujunkang, The director of microecological pharmaceutical research, Third Military Medical University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: liujunkang; dongying (Other Grant/Funding Number: Dongying leader pharmaceutical co.,LTD)
Record Dates: First submitted 2013-06-06; First posted 2013-07-09 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: diarrhea; abdominal pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Abdominal Pain | interventions — Acetylglucosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Starch capsule (Placebo Comparator): During the two weeks screening phase of the study, the daily dose of 3 tablets will be taken before breakfast, lunch and supper.
  Interventions: Drug: placebo
- N-acetyl-D-glucosamine (Experimental): During the 8-week treatment phase of the study,the dose of 100mg(3 tablets)per day will be taken.
  Interventions: Drug: N-acetyl-D-glucosamine

INTERVENTIONS:
Drug: N-acetyl-D-glucosamine
  Other Names: Atysamine (ATSM)
  Arms: N-acetyl-D-glucosamine
Drug: placebo
  Arms: Starch capsule

SUMMARY:
This study is a withdrawal randomized clinical trail to evaluate the clinical efficacy and safety of 1.1 chemical drugs N-acetyl glucosamine on Chinese IBS-D patients coming from four centers in chongqing. 180 IBS-D patients in this research are accord with the Rome III diagnostic criteria, screening/import period pain intensity scores of the NRS week mean value are 3.0 plus and the days which at least more than one time a stool type are 6 or 7 type over 2 days/week. Test cycle includes screening/import period (2 weeks), open treatment period (8 weeks), a double-blind placebo-controlled randomized withdrawal period (8 weeks), the main outcome measures are pain intensity (NRS score 11 point scale) and stool type ( Bristol type). And secondary endpoints included overall symptoms sensory scores, defecation frequency, abdominal distension, mucous stool and quality of life parameters (IBS-36 scale). After the end of the treatment period, the participants whose pain intensity and stool type are effective subjects into a randomized withdrawal period, analysis and comparison of the difference between treatment group and placebo group withdrawal rate and curative effect index score reduces.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, aged 18 to 65 years, inclusive.
* Based on the Roman III diagnostic criteria for diagnosis of IBS-D subjects, recurrent abdominal pain or discomfort (hard to describe the discomfort of pain), monthly attack within the past 3months at least 3 days. With two or more of the following three kinds of symptoms:

At least a portion of the time abdominal pain or defecate increase when discomfort.

At least a portion of the time abdominal pain or the row of loose stools when discomfort.

At least a portion of the time abdominal pain or discomfort improved after defecation.

Symptoms for at least 6 months before diagnosis

* Screening/import period pain intensity scores of the NRS week mean value are 3.0 plus and the days which at least more than one time a stool type are 6 or 7 type over 2 days/week.
* Voluntarily signed the informed consent form

Exclusion Criteria:

* The absorption of any known adverse
* History of gastrointestinal surgery ( not including appendectomy)
* History of organic gastrointestinal diseases: IBS, cancer etc.
* History of chronic diseases: anemia (hemoglobin<90g/L), pulmonary tuberculosis, diabetes or cardiovascular, liver, kidney, brain, and hematopoietic system and other serious diseases and psychiatric patients, AST(aspartate aminotransferase), ALT (alanine aminotransferase)> 1.5 times, BUN (blood urea nitrogen)> 1.2 times, Cr > 1.0 times normal.
* The disease of lactose intolerance, gallstones, endometriosis, easily confused with IBS symptoms of ;
* Progressive weight loss;
* Concomitant medication is unable to stop but affect the gastrointestinal movement and function in the experiment, such as antibiotic drugs, the drugs of regulating the intestinal microecology;
* Concomitant medication use continuously for more than a week but affect the gastrointestinal movement and function in the experiment, such as parasympathetic inhibitors, nondepolarizing agent, antidiarrheal, opioid formulation, etc;
* Other researchers think not suitable for the list;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Abdominal Pain Intensity | one and a half years
  As measured by numerical rating scale
Stool Consistency | one and a half years
  As measured by Bristol ' s scale

SECONDARY OUTCOMES:
General symptoms feel grading | one and a half years
  As measure by patient reported outcome measures
defecation frequency | one and a half years
  As measure by patient reported outcome measures
abdominal distension | one and a half years
  As measure by patient reported outcome measures
mucous stool | one and a half years
  As measure by patient reported outcome measures
life quality parameters | one and a half years
  As measure by healthy survey, SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Junkang Liu, Doctor, Study Chair — Third MMU
Locations (1):
- Daping hospital, Chongqing, Chongqing Municipality, China